CLINICAL TRIAL: NCT07210177
Title: Clinical and Radiographic Evaluation of Root Canal Treatments Performed Using Two Different Intracanal Medicaments
Brief Title: The Success of Root Canal Treatments Performed Using Two Different Intracanal Medicaments
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Seniha Miçooğulları Kurt, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUDF-ETK-24-6/7
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Root Canal Treatment; Intracanal Medicament; Post Operative Pain; Apical Periodontitis
Keywords: root canal treatment; chronic apical periodontitis; post operative pain; intracanal medicament
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two visit root canal treatment with Bio-C TEMP (Active Comparator): Two-visit root canal treatment will be performed on the study teeth. Bio-C TEMP (Angelus, Paraná, Brazil), a bioceramic-based intracanal medicament, will be placed in the root canals between appointments according to the manufacturer's instructions.
  Interventions: Other: Bio-C Temp Intracanal Medication
- Two visit root canal treatment with Meta Paste (Active Comparator): Two-visit root canal treatment will be performed on the study teeth. Meta Paste(Meta Biomed Co., Ltd., Chungcheongbuk-do, Korea) a calcium hydroxide based intracanal medicament, will be placed in theroot canals between appointments according to the manufacturer's instructions.
  Interventions: Other: Metapaste Intracanal Medication

INTERVENTIONS:
Other: Bio-C Temp Intracanal Medication — Bio-C Temp (Angelus, Paraná, Brazil) is a ready-to-use calcium silicate-based material designed for use between appointments. Bio-C Temp is indicated for use as a substitute for calcium hydroxide, as a medicament for necrotic teeth or root canal resurfacing treatments, and for the treatment of internal and external root resorption and immature teeth.
  Arms: Two visit root canal treatment with Bio-C TEMP
Other: Metapaste Intracanal Medication — Metapaste (Meta Bıomed Co.,Ltd., Chungcheongbuk-do,Korea) is a ready-to-use calcium hydroxide-based material designed for use between appointments.Metapaste is indicated for use as a medicament for necrotic teeth or root canal resurfacing treatments, and for the treatment of internal and external root resorption and immature teeth.
  Arms: Two visit root canal treatment with Meta Paste

SUMMARY:
Previously untreated, asymptomatic, single-rooted maxillary anterior teeth with periapical lesions <5 mm, no fractures, resorption, calcification, or recent antibiotic use will performed two-visit root canal treatment. Initial radiographs will be taken. After rubber-dam isolation, working length will be determined; canals prepared step-back to size #40 with sodium hypochlorite (NaOCl) irrigation, rinsed and dried. Between appointments, Metapaste or Bio-C TEMP will be placed as intracanal medicament for 7-10 days. At the second appointment medicaments removed, final irrigation performed and root canals obturated and restored. Pain scores recorded at 6h,12h,1d,2d,3d,4d,5d,6d,7d ; follow-ups at 6, 12 and 24 months.

DETAILED DESCRIPTION:
Within the scope of the project, two-visit root canal treatment will be performed on previously untreated, asymptomatic, single-rooted, single-canaled maxillary anterior teeth that have periapical lesions smaller than 5 mm on radiographs, no fractures or cracks, no internal or external resorption, no canal calcification, and no antibiotic use within the last week.

At the start of treatment, an initialradiograph will be taken of the tooth using a parallel film holder and archived. After rubber dam isolation, an access cavity will be prepared (all previous restorations will be removed if present). Working length will be determined by an apex locator. Root canal preparation will be performed using the step-back technique, with apical enlargement to at least size #40. Continuous irrigation with 2.5% NaOCl will be performed between each file. After instrumentation, the root canals will be rinsed with distilled water and dried with paper points.

Between appointments, to achieve additional disinfection of the root canals, Metapaste containing Ca(OH)₂ intracanal medicament (Meta Biomed Co., Ltd., Chungcheongbuk-do, Korea) and the bioceramic-based intracanal medicament Bio-C TEMP (Angelus, Paraná, Brazil) will be placed in the root canals according to the manufacturers' instructions. The intracanal distribution of the medicaments will be checked visually and radiographically, and the medicaments will be left in place for 7-10 days. Patients will be instructed on how to record their pain scores on the NRS scale and will be provided with contact information in case of any swelling or pain.

At the second appointment, after removal of the medicaments, a periapical radiograph will be taken for gutta-percha trial and verified according to the working length. In the final irrigation procedure, 5 mL of 17% ethylenediaminetetraacetic acid (EDTA), 5 mL of 2.5% NaOCl, distilled water and 2% chlorhexidine will be used respectively. After drying the root canals with paper points, they will be obturated with gutta-percha and a resin-based sealer using the cold lateral compaction technique, and the access cavities will be restored with composite resin. A final radiograph will be taken using the parallel technique with a parallel film holder.

Patients will again be given the NRS form and asked to return the completed forms after 7 days. Clinical follow-ups will be performed at the 6th, 12th, and 24th months, and follow-up radiographs will be taken using a parallel film holder. Changes in the size of the periapical lesions compared to baseline will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* with a non-contributory medical history, mature maxillary incisor teeth with periapical lesions, diagnosed as asymptomatic apical periodontitis

Exclusion Criteria:

* clinical symptoms, drainage, more than 5 mm loss of periodontal attachment, Teeth with periapical lesions larger than 5 mm previous endodontic treatment, non-restorable tooth patient with taken antibiotic or analgesics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain | Immediately after treatment, between appointments and after obturation for up to 7 days postoperatively
  Following two -visit root canal treatment performed with different intracanal medicament types , the Numerical Rating Scale (NRS) was used to assess both inter-appointment and after obturation. Compare the patients' pain levels, and the patients were instructed to record their pain at 6, 12, 24, 48, and 72 hours, as well as on the 7th day. Patients were informed that a score of 0 represented no pain, while a score of 10 represented the maximum pain, with higher scores indicating greater pain intensity

SECONDARY OUTCOMES:
Changes in the size and the PAI score of the periapical lesion | At 6,12 and 24 months after treatment.
  The rate of radiographic healing of the periapical lesion. Follow-up visits were performed for all patients in order to evaluate radiographic status. Changes in apical bone density indicating radiographic healing was assessed using Periapical Index (PAI) as the scoring system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No